CLINICAL TRIAL: NCT00263666
Title: A Phase II, Double-blind, Randomized, Placebo-controlled Study to Assess the Safety, Reactogenicity and Immunogenicity of Three Doses of GlaxoSmithKline (GSK) Biologicals' Oral Live Attenuated Human Rotavirus (HRV) Vaccine
Brief Title: A Study of Safety, Reactogenicity and Immunogenicity of HRV Vaccine in HIV Infected Infants in South Africa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 444563/022; 2015-001484-39 (EudraCT Number)
Record Dates: First submitted 2005-12-08; First posted 2005-12-09 (Estimated); Results first posted 2009-03-13 (Estimated); Last update posted 2020-11-23 (Actual); Status verified 2020-10

CONDITIONS: Infections, Rotavirus
MeSH Terms: conditions — Rotavirus Infections | interventions — RIX4414 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study was conducted in a double-blind manner. The parents/guardians of the subjects and the study personnel were unaware of the administered treatment (HRV vaccine or placebo).

ARMS (2):
- Rotarix Group (Experimental): Subjects received 3 doses of Rotarix vaccine co-administered with routine Tritanrix HepB Hib and Polio Sabin vaccines.
  Interventions: Biological: Rotarix; Biological: Tritanrix-HB+Hib; Biological: Polio Sabin
- Placebo Group (Placebo Comparator): Subjects received 3 doses of placebo co-administered with routine Tritanrix HepB Hib and Polio Sabin vaccines.
  Interventions: Biological: Placebo; Biological: Tritanrix-HB+Hib; Biological: Polio Sabin

INTERVENTIONS:
Biological: Rotarix — Oral vaccination
  Arms: Rotarix Group
Biological: Placebo — Oral administration
  Arms: Placebo Group
Biological: Tritanrix-HB+Hib — Concomitant routine vaccination, IM administration
Biological: Polio Sabin — Oral administration, concomitant routine vaccination

SUMMARY:
The aim of this study is to evaluate the reactogenicity, safety and immunogenicity of GSK Biologicals' human rotavirus (HRV) vaccine given concomitantly with routine vaccines including OPV in HIV positive infants. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

DETAILED DESCRIPTION:
HIV infected infants as determined prior to study entry (screening) and asymptomatic or mildly symptomatic (WHO stages I and II) of disease will be enrolled. The study will have two groups: Group HRV and Group Placebo. Three-dose immunisation will be administered at approximately 6, 10, and 14 weeks of age. Routine EPI (Expanded Program on Immunisation) vaccinations will be administered concomitantly with the study vaccines. At the time of first dose, subjects will be aged 6 to 10 weeks. This study will evaluate safety, reactogenicity and immunogenicity of the HRV vaccine relative to the placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/guardians can and will comply with the requirements of the protocol should be enrolled in the study.
* A male or female between, and including 6 and 10 weeks of age at the time of the first vaccination.
* Written informed consent obtained from the parents or guardians of the subject
* Documented HIV status of the subject as confirmed by PCR.
* HIV asymptomatic and HIV mildly symptomatic; Stages I and II disease according to WHO's most recent classification for HIV stages in infants and children.
* Born after a gestation period of 36 to 42 weeks.

Exclusion Criteria:

* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Previous routine vaccination except OPV, BCG and HBV vaccination at birth
* Any clinically significant history of chronic gastrointestinal disease including any uncorrected congenital malformation of the GI tract or other serious medical condition as determined by the investigator.
* History of allergic disease or reaction likely to be exacerbated by any component of the vaccine.
* Acute disease at time of enrolment.
* Gastroenteritis within 7 days preceding the study vaccine administration.
* Previous confirmed occurrence of RV gastroenteritis.
* Other conditions which in the opinion of the investigator may potentially interfere with interpretation of study outcomes.
* HIV moderately and severely symptomatic: stages III and IV according to WHO's recent classification.
* Administration of immunoglobulins and/or blood products since birth or planned administration during the study period.

Ages: 6 Weeks to 10 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2005-03-16 (Actual); Primary Completion 2008-02-07 (Actual); Study Completion 2008-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- South Africa (6):
  - GSK Investigational Site, Attridgerville, Gauteng
  - GSK Investigational Site, Coronationville, Gauteng
  - GSK Investigational Site, Garankuwa, North West
  - GSK Investigational Site, Brits
  - GSK Investigational Site, Capital Park
  - GSK Investigational Site, Ga-Rankuwa

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Buyse H, Vinals C, Karkada N, Han HH. The human rotavirus vaccine Rotarix in infants: an integrated analysis of safety and reactogenicity. Hum Vaccin Immunother. 2014;10(1):19-24. doi: 10.4161/hv.26476. Epub 2013 Oct 8. PMID 24047799
- [Background] Steele AD, Madhi SA, Louw CE, Bos P, Tumbo JM, Werner CM, Bicer C, De Vos B, Delem A, Han HH. Safety, Reactogenicity, and Immunogenicity of Human Rotavirus Vaccine RIX4414 in Human Immunodeficiency Virus-positive Infants in South Africa. Pediatr Infect Dis J. 2011 Feb;30(2):125-30. doi: 10.1097/INF.0b013e3181f42db9. PMID 20842070
- [Derived] Ruiz-Palacios GM, Perez-Schael I, Velazquez FR, Abate H, Breuer T, Clemens SC, Cheuvart B, Espinoza F, Gillard P, Innis BL, Cervantes Y, Linhares AC, Lopez P, Macias-Parra M, Ortega-Barria E, Richardson V, Rivera-Medina DM, Rivera L, Salinas B, Pavia-Ruz N, Salmeron J, Ruttimann R, Tinoco JC, Rubio P, Nunez E, Guerrero ML, Yarzabal JP, Damaso S, Tornieporth N, Saez-Llorens X, Vergara RF, Vesikari T, Bouckenooghe A, Clemens R, De Vos B, O'Ryan M; Human Rotavirus Vaccine Study Group. Safety and efficacy of an attenuated vaccine against severe rotavirus gastroenteritis. N Engl J Med. 2006 Jan 5;354(1):11-22. doi: 10.1056/NEJMoa052434. PMID 16394298
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 444563/022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 444563/022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 444563/022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 444563/022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 444563/022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 444563/022 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In case of discrepancy between the HIV results (DNA PCR positive, viral load negative), performed at the Screening Visit (one week prior to first vaccination) the infants were not enrolled in the study.
Period: Overall Study
Arm/Group | Rotarix Group | Placebo Group
Started | 50 | 50
Completed | 43 | 39
Not Completed | 7 | 11
Not completed — Adverse Event | 6 | 8
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rotarix Group | Placebo Group | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 7.1 (1.10) | 6.9 (1.02) | 7.0 (1.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 25 | 53
  Male | 22 | 25 | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Grade "2" or Grade "3" Fever, Vomiting or Diarrhea
Description: Symptoms reported in the table include: Fever: temperature (axillary route) > 38.0 degree Celsius (°C); Diarrhea: ≥ 4 looser than normal stools/day; Vomiting: ≥ 2 episodes of vomiting/day.
Time Frame: Within the 15-day solicited follow-up period after any dose
Population: The analysis was performed on the Total Vaccinated Cohort which included the vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 50 | 50
Participants | 26 | 28

2. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Symptoms
Description: An unsolicited symptom was any spontaneously reported untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Within 30 days after any dose
Population: Analysis was performed on the Total Vaccinated Cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 50 | 50
Participants | 47 | 48

3. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events
Description: A serious adverse event (SAE) is any untoward medical occurrence that: results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject, or may evolve into one of the outcomes listed above.
Time Frame: Until 2 months after dose 3 (for subjects RV negative at Day 42 post-dose 3) or until end of RV shedding (for subjects who shed RV at Day 42 post-dose 3)
Population: Analysis was performed on the Total Vaccinated Cohort.
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 50 | 50
Participants | 17 | 12

4. Secondary Outcome: Number of Subjects Reporting Each Type of Solicited Symptom
Description: Solicited symptoms included Cough, Diarrhea (3 or more looser than normal stools/day), Fever (axillary temperature ≥ 37.5°C), Irritability, Loss of appetite, and Vomiting.
Time Frame: Within the 15-day solicited follow-up period after each dose
Population: Analysis was performed on the Total Vaccinated Cohort, which included vaccinated subjects for whom data were available and who had their symptom sheets completed.
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 50 | 50
Participants
  Cough, after dose 1 | 24 | 25
  Diarrhoea, after dose 1 | 8 | 8
  Fever, after dose 1 | 20 | 19
  Irritability, after dose 1 | 24 | 24
  Loss of appetite, after dose 1 | 18 | 19
  Vomiting, after dose 1 | 11 | 10
  Cough, after dose 2: number analyzed (Participants) | 46 | 48
  Cough, after dose 2 | 18 | 19
  Diarrhoea, after dose 2: number analyzed (Participants) | 46 | 48
  Diarrhoea, after dose 2 | 3 | 7
  Fever, after dose 2: number analyzed (Participants) | 46 | 48
  Fever, after dose 2 | 15 | 12
  Irritability, after dose 2: number analyzed (Participants) | 46 | 48
  Irritability, after dose 2 | 20 | 19
  Loss of appetite, after dose 2: number analyzed (Participants) | 46 | 48
  Loss of appetite, after dose 2 | 15 | 15
  Vomiting, after dose 2: number analyzed (Participants) | 46 | 48
  Vomiting, after dose 2 | 9 | 10
  Cough, after dose 3: number analyzed (Participants) | 45 | 44
  Cough, after dose 3 | 18 | 17
  Diarrhoea, after dose 3: number analyzed (Participants) | 45 | 44
  Diarrhoea, after dose 3 | 7 | 4
  Fever, after dose 3: number analyzed (Participants) | 45 | 44
  Fever, after dose 3 | 17 | 13
  Irritability, after dose 3: number analyzed (Participants) | 45 | 44
  Irritability, after dose 3 | 17 | 18
  Loss of appetite, after dose 3: number analyzed (Participants) | 45 | 44
  Loss of appetite, after dose 3 | 10 | 12
  Vomiting, after dose 3: number analyzed (Participants) | 45 | 44
  Vomiting, after dose 3 | 12 | 6

5. Secondary Outcome: The Number of Subjects With no Evidence of Immunosuppression and Moderate/ Severe Suppression, Based on CD4+ Absolute Cell Count and CD4+ Percent
Description: Severe suppression: CD4+ cells/microliter (μl) < 750 and CD4+ percent < 15 percent (%); No evidence of suppression: CD4+ cells/μl ≥ 1500 and CD4+ percent ≥ 25%; Moderate suppression = all other CD4+ cell count and CD4+ % combinations.
Time Frame: At the screening visit and 2 months after dose 3 (Visit 4)
Population: Analysis was performed on the Total Vaccinated Cohort, which included vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 50 | 50
Participants
  Severe suppression at screening | 1 | 2
  Moderate suppression at screening | 12 | 15
  No suppression at screening | 37 | 33
  Severe suppression at Visit 4: number analyzed (Participants) | 43 | 39
  Severe suppression at Visit 4 | 11 | 7
  Moderate suppression at Visit 4: number analyzed (Participants) | 43 | 39
  Moderate suppression at Visit 4 | 15 | 18
  No suppression at Visit 4: number analyzed (Participants) | 43 | 39
  No suppression at Visit 4 | 13 | 10
  Unknown at Visit 4: number analyzed (Participants) | 43 | 39
  Unknown at Visit 4 | 4 | 4

6. Secondary Outcome: Human Immunodeficiency Virus (HIV) Viral Load
Description: The HIV viral load was expressed as mean and standard deviation of the base-10 logarithm of HIV-1 ribonucleic acid (RNA) copies per milliliter (mL).
Time Frame: At the screening visit and 2 months after dose 3
Population: Analysis was performed on the Total Vaccinated Cohort, which included vaccinated subjects for whom data were available.
Measure: Mean (Standard Deviation); unit: base-10 logarithm of copies/milliliter
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 50 | 50
base-10 logarithm of copies/milliliter
  At screening | 5.7 (0.52) | 5.7 (0.51)
  Two months after dose 3: number analyzed (Participants) | 43 | 36
  Two months after dose 3 | 5.6 (0.77) | 5.7 (0.51)

7. Secondary Outcome: Number of Subjects Who Seroconverted Against Rotavirus
Description: A subject with anti-rotavirus Immunoglobulin (IgA) antibody concentration < 20 units/milliliter (U/mL) before vaccination and ≥ 20 U/mL after vaccination is considered as seroconverted.
Time Frame: Two months after dose 3
Population: Analysis was performed on subjects from the According to Protocol Cohort for immunogenicity for whom results were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 21 | 22
Participants | 12 | 4

8. Secondary Outcome: Number of Subjects With Vaccine Take
Description: Vaccine take: appearance of serum IgA to rotavirus at a concentration of ≥ 20 U/ml or rotavirus shedding in any stool sample collected from the Screening Visit to 2 months after dose 3 for subjects initially negative for rotavirus.
Time Frame: Two months after dose 3
Population: Analysis was performed on subjects from the According To Protocol Cohort for immunogenicity for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 23 | 22
Participants | 15 | 7

9. Secondary Outcome: Serum Rotavirus Immunoglobulin A (IgA) Antibody Concentrations
Description: Concentrations are given as geometric mean concentrations (GMC) for anti-rotavirus IgA antibodies.
Time Frame: Two months after dose 3
Population: The analysis was performed on the According To Protocol Cohort for immunogenicity for whom data were available. In the Placebo group, GMCs were all < 20 U/ml, hence values were not computed.
Measure: Geometric Mean (95% Confidence Interval); unit: Units/milliliter
Arm/Group | Rotarix Group
Number analyzed (Participants) | 21
Units/milliliter | 75.5 [29.1 to 195.7]

10. Secondary Outcome: Number of Subjects With Anti-polyribosyl Ribitol Phosphate (PRP) Antibody Concentrations More Than or Equal to the Cut-off Value
Description: Cut-off values for anti-PRP antibody concentrations were ≥ 0.15 and ≥ 1.0 microgram/milliliter (µg/mL).
Time Frame: Two months after dose 3
Population: The analysis was performed on the According To Protocol Cohort for immunogenicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 25 | 24
Participants
  ≥ 0.15 µg/mL | 20 | 23
  ≥ 1 µg/mL | 20 | 22

11. Secondary Outcome: Geometric Mean Concentration for Anti-PRP Antibodies
Description: Anti-PRP antibody concentrations are presented as geometric mean concentrations, expressed in microgram/milliliter (μg/mL).
Time Frame: Two months after dose 3
Population: The analysis was performed on the According to Protocol cohort for immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: microgram/milliliter
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 25 | 24
microgram/milliliter | 4.641 [1.764 to 12.215] | 4.865 [2.322 to 10.192]

12. Secondary Outcome: Number of Subjects With Anti-diphtheria and Anti-tetanus Toxoids Antibody Concentrations More Than or Equal to the Cut-off Value
Description: The cut-off value was ≥ 0.1 International Units/milliliter (IU/mL).
Time Frame: Two months after dose 3
Population: The analysis was performed on the According To Protocol cohort for immunogenicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 25 | 25
Participants
  Anti-diphtheria | 19 | 19
  Anti-tetanus | 23 | 24

13. Secondary Outcome: Geometric Mean Concentration for Anti-diphtheria and Anti-tetanus Toxoids Antibodies
Description: Anti-diphteria and anti-tetanus toxoids antibody concentrations are presented as geometric mean concentrations, expressed in international units/milliliter (IU/mL).
Time Frame: Two months after dose 3
Population: The analysis was performed on the According to Protocol cohort for immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: International Units / milliliter
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 25 | 25
International Units / milliliter
  Anti-tetanus | 1.457 [0.794 to 2.674] | 1.035 [0.647 to 1.656]
  Anti-diphtheria | 0.283 [0.167 to 0.481] | 0.219 [0.143 to 0.337]

14. Secondary Outcome: Number of Subjects With Anti-hepatitis B (HBs) Antibody Concentrations More Than or Equal to the Cut-off Value
Description: The cut-off value was ≥ 10 milli international units/milliliter (mIU/mL).
Time Frame: Two months after dose 3
Population: The analysis was performed on the According To Protocol cohort for immunogenicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 23 | 20
Participants | 15 | 11

15. Secondary Outcome: Geometric Mean Concentration for Anti-HBs Antibodies
Description: Anti-HBs antibody concentrations are presented as geometric mean concentrations, expressed in milli international units/milliliter (mIU/mL).
Time Frame: Two months after dose 3
Population: The analysis was performed on the According to Protocol cohort for immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: Milli International Units/milliliter
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 23 | 20
Milli International Units/milliliter | 25.6 [14.3 to 45.8] | 18.9 [9.9 to 36.1]

16. Secondary Outcome: Number of Subjects With Anti-Bordetella Pertussis (BPT) Antibody Concentrations More Than or Equal to the Cut-off Value
Description: The cut-off value was ≥ 15 Enzyme Linked Immunosorbent Assay Unit/milliliter (EL.U/mL).
Time Frame: Two months after dose 3
Population: The analysis was performed on the According To Protocol cohort for immunogenicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 25 | 24
Participants | 19 | 14

17. Secondary Outcome: Geometric Mean Concentration for Anti-BPT Antibodies
Description: Anti-BPT antibody concentrations are presented as geometric mean concentrations, expressed in ELISA units/milliliter (EL.U/mL).
Time Frame: Two months after dose 3
Population: The analysis was performed on the According to Protocol cohort for immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA-Units/milliliter
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 25 | 24
ELISA-Units/milliliter | 28.8 [19.3 to 42.8] | 18.1 [12.8 to 25.6]

18. Secondary Outcome: Number of Subjects With Anti-polio Types 1, 2 and 3 Antibody Titers More Than or Equal to the Cut-off Value
Description: The cut-off value was ≥ 1:8. The lowest dilution at which serum samples were tested was 1:8, from which a test was considered positive.
Time Frame: Two months after dose 3
Population: The analysis was performed on the According To Protocol cohort for immunogenicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 25 | 24
Participants
  Anti-polio type 1 | 19 | 15
  Anti-polio type 2 | 23 | 21
  Anti-polio type 3: number analyzed (Participants) | 25 | 23
  Anti-polio type 3 | 18 | 15

19. Secondary Outcome: Geometric Mean Titer for Anti-polio Types 1, 2 and 3 Antibodies.
Description: Anti-polio types 1, 2 and 3 antibody titers are presented as geometric mean titers.
Time Frame: Two months after dose 3
Population: The analysis was performed on the According To Protocol cohort for immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 25 | 24
Titer
  Anti-polio 1 | 90.5 [36.4 to 225.3] | 53.0 [19.4 to 144.5]
  Anti-polio 2 | 142.6 [60.8 to 334.2] | 252.4 [91.2 to 698.7]
  Anti-polio 3: number analyzed (Participants) | 25 | 23
  Anti-polio 3 | 44.7 [19.2 to 104.2] | 66.0 [22.6 to 192.2]

20. Secondary Outcome: Rotavirus Antigen Excretion in Stool Samples
Description: Number of subjects with rotavirus detected by Enzyme Linked Immunosorbent Assay (ELISA) in stool samples collected from Dose 1 until study end.
Time Frame: At day of each vaccination and at planned days following each vaccine dose until 2 months after dose 3 or until end of RV shedding
Population: The analysis was performed on the According to Protocol Cohort for immunogenicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 25 | 25
Participants | 11 | 5

21. Secondary Outcome: Rotavirus in Diarrheal Stool Samples
Description: Number of subjects reporting at least one rotavirus (vaccine strain or wild type rotavirus) gastroenteritis episode.
Time Frame: From Dose 1 until 2 months after dose 3 or until end of RV shedding
Population: Analysis was performed on the Total Vaccinated Cohort
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 50 | 50
Participants | 4 | 4

22. Secondary Outcome: Rotavirus Vaccine Strain Identification
Description: Number of gastroenteritis (GE) episodes classified by rotavirus vaccine strain/serotype. Unknown: These samples were typed post hoc and found "G1P8" vaccine type for one subject in HRV group, "G3P8" and "G2P4" for subjects in placebo group.
Time Frame: From dose 1 until 2 months after dose 3 or until end of RV shedding
Population: Analysis was performed on the Total Vaccinated Cohort.
Measure: Number; unit: Number of episodes
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 50 | 50
Number of episodes
  G1WT+P8WT | 2 | 0
  G2+P4 | 0 | 1
  G3+P8 | 0 | 1
  GX+P6 | 1 | 0
  Unknown | 1 | 2

23. Secondary Outcome: Enteric Pathogens Identification
Description: Number of subjects reporting gastroenteritis (GE) episodes classified by enteric pathogen tests results.
Time Frame: From Dose 1 until 2 months after dose 3 or until end of RV shedding
Population: The analysis was performed on the subjects from the Total Vaccinated Cohort with gastroenteritis episodes reported between the first dose and the last visit and for whom stools were collected.
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 29 | 34
Participants
  Campylobacter, negative | 18 | 24
  Campylobacter, positive | 0 | 0
  Campylobacter, unknown | 11 | 10
  E. histolytica, negative | 18 | 24
  E. histolytica, positive | 0 | 0
  E. histolytica, unknown | 11 | 10
  Salmonella, negative | 17 | 24
  Salmonella, positive | 1 | 0
  Salmonella, unknown | 11 | 10
  Sto Epec, negative | 3 | 5
  Sto Epec, positive | 0 | 0
  Sto Epec, unknown | 26 | 29
  Sto G.Lamblia, negative | 18 | 24
  Sto G.Lamblia, positive | 0 | 0
  Sto G.Lamblia, unknown | 11 | 10
  Sto Shigella, negative | 18 | 24
  Sto Shigella, positive | 0 | 0
  Sto Shigella, unknown | 11 | 10
  Sto Yersinia, negative | 18 | 24
  Sto Yersinia, positive | 0 | 0
  Sto Yersinia, unknown | 11 | 10

24. Secondary Outcome: Number of Subjects With the RV in Stool Samples
Description: Number of subjects with presence of RV in stool samples (shedding) collected at pre-determined time points by RV type (Yes, No, Mixed type = G1V+G1WT+G2+G3+P4+P8V+P8WT and results not available [NA]).
Time Frame: From Dose 1 until post Dose 3
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Rotarix Group | Placebo Group
Number analyzed (Participants) | 26 | 7
Participants
  Dose 1 (Day 7; Yes ): number analyzed (Participants) | 9 | 1
  Dose 1 (Day 7; Yes ) | 7 | 0
  Dose 1 (Day 7; No): number analyzed (Participants) | 9 | 1
  Dose 1 (Day 7; No) | 0 | 0
  Dose 1 (Day 7; NA): number analyzed (Participants) | 9 | 1
  Dose 1 (Day 7; NA) | 2 | 1
  Dose 1 (Day 14; Yes): number analyzed (Participants) | 4 | 2
  Dose 1 (Day 14; Yes) | 0 | 0
  Dose 1 (Day 14; No): number analyzed (Participants) | 4 | 2
  Dose 1 (Day 14; No) | 0 | 1
  Dose 1 (Day 14; Mixed): number analyzed (Participants) | 4 | 2
  Dose 1 (Day 14; Mixed) | 0 | 1
  Dose 1 (Day 14; NA): number analyzed (Participants) | 4 | 2
  Dose 1 (Day 14; NA) | 4 | 0
  Dose 1 (Day 21; Yes): number analyzed (Participants) | 5 | 1
  Dose 1 (Day 21; Yes) | 1 | 0
  Dose 1 (Day 21; No): number analyzed (Participants) | 5 | 1
  Dose 1 (Day 21; No) | 0 | 1
  Dose 1 (Day 21; NA): number analyzed (Participants) | 5 | 1
  Dose 1 (Day 21; NA) | 4 | 0
  Dose 2 (Day 7; Yes): number analyzed (Participants) | 0 | 1
  Dose 2 (Day 7; Yes) |  | 0
  Dose 2 (Day 7; No): number analyzed (Participants) | 0 | 1
  Dose 2 (Day 7; No) |  | 1
  Dose 2 (Day 7; NA): number analyzed (Participants) | 0 | 1
  Dose 2 (Day 7; NA) |  | 0
  Dose 2 (Day 14; Yes): number analyzed (Participants) | 1 | 0
  Dose 2 (Day 14; Yes) | 0 |
  Dose 2 (Day 14; No): number analyzed (Participants) | 1 | 0
  Dose 2 (Day 14; No) | 0 |
  Dose 2 (Day 14; NA): number analyzed (Participants) | 1 | 0
  Dose 2 (Day 14; NA) | 1 |
  Dose 2 (Day 21; Yes): number analyzed (Participants) | 2 | 0
  Dose 2 (Day 21; Yes) | 0 |
  Dose 2 (Day 21; No): number analyzed (Participants) | 2 | 0
  Dose 2 (Day 21; No) | 0 |
  Dose 2 (Day 21; NA): number analyzed (Participants) | 2 | 0
  Dose 2 (Day 21; NA) | 2 |
  Dose 3 (Day 7; Yes): number analyzed (Participants) | 1 | 1
  Dose 3 (Day 7; Yes) | 0 | 0
  Dose 3 (Day 7; No): number analyzed (Participants) | 1 | 1
  Dose 3 (Day 7; No) | 0 | 1
  Dose 3 (Day 7; NA): number analyzed (Participants) | 1 | 1
  Dose 3 (Day 7; NA) | 1 | 0
  Dose 3 (Day 14; Yes): number analyzed (Participants) | 2 | 0
  Dose 3 (Day 14; Yes) | 2 |
  Dose 3 (Day 14; No): number analyzed (Participants) | 2 | 0
  Dose 3 (Day 14; No) | 0 |
  Dose 3 (Day 14; NA): number analyzed (Participants) | 2 | 0
  Dose 3 (Day 14; NA) | 0 |
  Dose 3 (Day 42; Yes): number analyzed (Participants) | 1 | 1
  Dose 3 (Day 42; Yes) | 0 | 0
  Dose 3 (Day 42; No): number analyzed (Participants) | 1 | 1
  Dose 3 (Day 42; No) | 0 | 0
  Dose 3 (Day 42; NA): number analyzed (Participants) | 1 | 1
  Dose 3 (Day 42; NA) | 1 | 1
  Post Dose 3 (Day 0; Yes): number analyzed (Participants) | 1 | 0
  Post Dose 3 (Day 0; Yes) | 0 |
  Post Dose 3 (Day 0; No): number analyzed (Participants) | 1 | 0
  Post Dose 3 (Day 0; No) | 0 |
  Post Dose 3 (Day 0; NA): number analyzed (Participants) | 1 | 0
  Post Dose 3 (Day 0; NA) | 1 |
  Overall total (overall total; Yes) | 10 | 0
  Overall total (overall total; No) | 0 | 4
  Overall total (overall total; Mixed type) | 0 | 1
  Overall total (overall total; NA) | 16 | 2

ADVERSE EVENTS:
Time Frame: Solicited general symptoms during the 15-day (Days 0-14) post-vaccination period following each dose and across doses, unsolicited AEs within 31 days (Days 0-30) after any vaccination and SAEs throughout the study period.
Arm/Group | Rotarix Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 6/50 | 9/50
Serious Adverse Events (participants affected / at risk) | 17/50 | 12/50
Other Adverse Events (participants affected / at risk) | 48/50 | 47/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rotarix Group (N=50) | Placebo Group (N=50)
Anemia (Blood and lymphatic system disorders) | 1 | 1
Conjunctivitis (Eye disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Sudden infant death syndrome (General disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Bronchiolitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 7 | 4
Lobar pneumonia (Infections and infestations) | 0 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 2 | 2
Pneumonia (Infections and infestations) | 1 | 3
Lymph node tuberculosis (Infections and infestations) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 2 | 4
Tuberculosis (Infections and infestations) | 1 | 0
Dysentery (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 6 | 3
HIV infection (Infections and infestations) | 1 | 0
Meningitis (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 2 | 0
Sepsis (Infections and infestations) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Marasmus (Metabolism and nutrition disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rotarix Group (N=50) | Placebo Group (N=50)
Lymphadenopathy (Blood and lymphatic system disorders) | 5 | 3
Splenomegaly (Blood and lymphatic system disorders) | 2 | 4
Constipation (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 1 | 5
Pyrexia (General disorders) | 3 | 6
Upper respiratory tract infection (Infections and infestations) | 18 | 14
Pulmonary tuberculosis (Infections and infestations) | 2 | 4
Influenza (Infections and infestations) | 6 | 0
Pharyngitis (Infections and infestations) | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 4 | 4
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 5 | 4
Eczema (Skin and subcutaneous tissue disorders) | 2 | 8
Rash (Skin and subcutaneous tissue disorders) | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 3
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 3
Weight decreased (Investigations) | 1 | 4
Cough (General disorders) | 35 | 31
Diarrhoea (General disorders) | 16 | 16
Fever (General disorders) | 30 | 28
Irritability (General disorders) | 31 | 28
Loss of appetite (General disorders) | 23 | 23
Vomiting (General disorders) | 19 | 15
Bronchopneumonia (Infections and infestations) | 11 | 6
Gastroenteritis (Infections and infestations) | 9 | 9
Oral candidiasis (Infections and infestations) | 15 | 19
Otitis media (Infections and infestations) | 4 | 6
Sepsis (Infections and infestations) | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.